CLINICAL TRIAL: NCT02162784
Title: An Open-Label, Randomized, Cross-Over Study to Evaluate the Dose Response of SYN006 HFA MDI in Asthma Patients
Brief Title: Efficacy Study of SYN006 HFA MDI in Asthma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intech Biopharm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INTB012; INTB012 (Other: Taiwan FDA)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Procaterol; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Budesonide/procaterol 180/10mcg X1 (Experimental): HFA MDI, oral inhalation, 180/10mcg, one puff
  Interventions: Drug: Budesonide/Procaterol, 180/10mcg X1
- Budesonide/Procaterol, 180/10mcg X2 (Experimental): HFA MDI, oral inhalation, two puffs
  Interventions: Drug: Budesonide/procaterol 180/10 mcg X 2
- Albuterol HFA MDI 100 mcg X2 (Active Comparator): HFA MDI, oral inhalation, 100mcg, two puffs
  Interventions: Drug: Albuterol HFA MDI 100mcg X2

INTERVENTIONS:
Drug: Budesonide/Procaterol, 180/10mcg X1 — one puff
  Other Names: Synbitide
  Arms: Budesonide/procaterol 180/10mcg X1
Drug: Budesonide/procaterol 180/10 mcg X 2 — 2 puffs
  Other Names: Synbitide
  Arms: Budesonide/Procaterol, 180/10mcg X2
Drug: Albuterol HFA MDI 100mcg X2 — HFA MDI, 100mcg, 2 puffs
  Other Names: Ventolin
  Arms: Albuterol HFA MDI 100 mcg X2

SUMMARY:
The objective of the study is to evaluate the dose response of SYN006 HFA MDI, which is a combination drug product of budesonide and procaterol hydrochloride, in asthma patients. Patients with mild to moderate asthma will be recruited. There will be two study medication administered in this study. The investigational medication is SYN006 (Budesonide/Procaterol hydrochloride, 180 mcg/10 mcg per inhalation) and the active comparative medication is Ventolin (Salbutamol sulfate 100 mcg per inhalation). The study medication will be administered by oral inhalation with the supervision of the investigator or a qualified staff.

DETAILED DESCRIPTION:
Three treatments will be administered in a patient:

* A. Two inhalations of Ventolin 100 mcg,
* B. One inhalation of SYN006 180/10 mcg,
* C. Two inhalations of SYN006 180/10 mcg.

Patients will be received the study treatment according to one of the six treatment sequences according to the randomization schedule:

1. A-B-C,
2. B-A-C,
3. C-A-B,
4. C-B-A,
5. A-C-B,
6. B-C-A.

The efficacy endpoint is

* The change in Forced Expiratory Volume in 1 second (FEV1) within 6 hours.
* The change in Peak Expiratory Flow Rate (PEFR) within 6 hours.
* The change in Force Vital Capacity (FVC) within 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged >= 16 years old
* History of FEV1 >=12% and 200 ml increase after inhalation of short-acting beta 2-agonist;
* Pre-bronchodilator FEV1 > 60% and < 90% of predicted normal value at enrollment;
* Ability to inhale correctly through MDI inhaler
* Written informed consent obtained.
* Diagnosis of mild to moderate persistent asthma according to GINA with a documented history of at least 6 months duration.

Mild Persistent:

1. Symptoms more than once a week but less than once a day
2. Nocturnal symptoms more than twice a month
3. Exacerbations may affect activity and sleep
4. FEV1 or PEF >= 80% predicted
5. PEF or FEV1 variability < 20 - 30%

Moderate Persistent:

1. Symptoms daily
2. Nocturnal symptoms more than once a week
3. Exacerbations may affect activity and sleep
4. Daily use of inhaled short-acting beta2-agonist
5. FEV1 or PEF > 60% - < 80% predicted
6. PEF or FEV1 variability > 30%

Exclusion Criteria:

* Currently uncontrolled asthma according to GINA guideline;
* Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients;
* Inability to carry out pulmonary function testing;
* Severe asthma associated with reduced lung function;
* Clinically significant or unstable concurrent diseases: uncontrolled hyperthyroidism, significant hepatic impairment, poorly controlled pulmonary disease (tuberculosis, active mycotic infection of the lung), gastrointestinal (e.g., active peptic ulcer), neurological or haematological autoimmune diseases;
* Abnormal ECG at enrollment;
* History of near-fatal asthma and/or admission intensive care unit because of asthma;
* History or current evidence of heart failure, coronary artery disease, myocardial infarction, severe hypertension, or cardiac arrhythmias;
* Percutaneous transluminal coronary angioplasty (PTCA) or coronary artery by-pass graft (CABG) during the previous 6 months at enrollment;
* Hospitalization for asthma during the past 3 months at enrollment;
* Evidence of severe asthma exacerbation or symptomatic infection of the airways in the previous 3 months at enrollment;
* Current smokers or recent (less than one year) ex-smokers, defined as smoking at least 10 pack/years;
* History of alcohol or drug abuse;
* Pregnant or lactating females or not able to exclude pregnancy during the study period;
* Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study;
* Patients who received any investigational new drug within the last 3 months at enrollment;
* Patients who have been previously enrolled in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The variation of study medications by the area under curve of FEV1 from 0 to 120 minutes (AUC0-120min ) after inhalation. | 5, 20, 40, 60, 90, 120 minutes, 4, and 6 hours after the inhalation

SECONDARY OUTCOMES:
The change in Forced Expiratory Volume in 1 second (FEV1) of study medication. | 5, 20, 40, 60, 90, 120 minutes, 4, and 6 hours after the inhalation
The change in Peak Expiratory Flow Rate (PEFR) of study medication. | 5, 20, 40, 60, 90, 120 minutes, 4, and 6 hours after the inhalation
The change in Forced Vital Capacity (FVC) of study medication. | 5, 20, 40, 60, 90, 120 minutes, 4, and 6 hours after the inhalation
The variation of study medications by the area under curve of PEFR from 0 to 120 minutes (AUC0-120min ) after inhalation. | 5, 20, 40, 60, 90, 120 minutes, 4, and 6 hours after the inhalation
The variation of study medications by the area under curve of FVC from 0 to 120 minutes (AUC0-120min ) after inhalation. | 5, 20, 40, 60, 90, 120 minutes, 4, and 6 hours after the inhalation

OTHER OUTCOMES:
Adverse events, vital signs, abnormal ECG outcome. | 5, 20, 40, 60, 90, 120 minutes, 4, and 6 hours after the inhalation

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei